CLINICAL TRIAL: NCT02544360
Title: Smokerface: A Photoaging Mobile App Promoting Poster Campaign for Preventing Smoking in Secondary Schools: Randomized Controlled Trial
Brief Title: A Photoaging Mobile App Promoting Poster Campaign for Preventing Smoking in Secondary Schools
Acronym: Smokerface
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Giessen (Other)
Collaborators: Heidelberg University (Other); Goethe University (Other); Massachusetts General Hospital (Other); Universität Duisburg-Essen (Other); Harvard University (Other); University Medical Center Goettingen (Other); University of Freiburg (Other); University of Bonn (Other); Technical University of Munich (Other); University of Homburg (Other); German Center for Lung Research (Other); The German Heart Foundation (Other)
Responsible Party: Principal Investigator, Titus J. Brinker, MD candidate, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 040890
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Tobacco Addiction; Smoking Related Diseases; Adolescent Smoking
Keywords: photoaging mobile apps; adolescent smoking; tobacco prevention; school-based prevention; adolescent health; school health; smoking; tobacco
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Schools in this arm receive a photoaging mobile app promoting poster campaign revealing the effects of smoking on the users face via a self portrait (i.e. a "selfie").
  Interventions: Behavioral: Photoaging mobile app promoting poster campaign.
- Control (No Intervention): The control group consists of schools participating in the survey but not receiving the intervention.

INTERVENTIONS:
Behavioral: Photoaging mobile app promoting poster campaign. — Schools in this arm receive a photoaging mobile app promoting poster campaign revealing the effects of smoking on the users face via a self portrait (i.e. a "selfie").
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether photoaging mobile app promoting poster campaigns are effective to reduce smoking prevalence among adolescents in Germany. This is measured via questionnaire.

DETAILED DESCRIPTION:
This RCT will investigate a novel mean of school-based tobacco prevention: Photoaging app promoting poster campaigns. The effects are measured via questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Students from Germany aged 9 to 14 years at baseline attending grades six and seven of regular German secondary schools (such as grammar, general, intermediate or comprehensive school) are eligible.

Exclusion Criteria:

* Older or younger pupils or pupils from other school types or countries or schools who previously participated in an event where the Smokerface app was presented are not eligible.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12000 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The change in smoking prevalence between baseline and 24 months of follow-up between the two groups measured via questionnaires. | 24 months post intervention
  The change in smoking prevalence between baseline and 24 months of follow-up between the two groups. A smoker is defined as someone who claims to have smoked cigarettes at least once in the past 30 days.

SECONDARY OUTCOMES:
Difference in attitude towards smoking between the two groups at 24 months follow-up measured via questionnaires. | 24 months post intervention
  Difference in attitude towards smoking between the two groups at 24 months follow-up.
The change in never-smokers between baseline and 24 months of follow-up between the two groups measured via questionnaires. | 24 months post intervention
  The change in never-smokers between baseline and 24 months of follow-up between the two groups measured via questionnaires.
The difference in the number of quitters (=cigarette smokers at baseline but not at endline) between baseline and 24 months of follow-up between the two groups measured via questionnaires. | 24 months post intervention
  The difference in the number of quitters (=quitters are participants who are cigarette smokers at baseline but not at endline) between baseline and 24 months of follow-up between the two groups measured via questionnaires.
The difference in the number of starters (=starters are participants who are not cigarette smokers at baseline but at endline) between baseline and 24 months of follow-up between the two groups measured via questionnaires. | 24 months post intervention
  The difference in the number of starters (=starters are participants who are not cigarette smokers at baseline but at endline) between baseline and 24 months of follow-up between the two groups measured via questionnaires.
The change in smoking prevalence between baseline and 24 months of follow-up between female participants of the two groups measured via questionnaires. | 24 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Titus J Brinker, Principal Investigator — University of Giessen
Locations (1):
- University of Gießen, Giessen, Hesse, Germany

REFERENCES:
- [Background] Brinker TJ, Seeger W. Photoaging Mobile Apps: A Novel Opportunity for Smoking Cessation? J Med Internet Res. 2015 Jul 27;17(7):e186. doi: 10.2196/jmir.4792. No abstract available. PMID 26215210
- [Derived] Brinker TJ, Holzapfel J, Baudson TG, Sies K, Jakob L, Baumert HM, Heckl M, Cirac A, Suhre JL, Mathes V, Fries FN, Spielmann H, Rigotti N, Seeger W, Herth F, Groneberg DA, Raupach T, Gall H, Bauer C, Marek P, Batra A, Harrison CH, Taha L, Owczarek A, Hofmann FJ, Thomas R, Mons U, Kreuter M. Photoaging smartphone app promoting poster campaign to reduce smoking prevalence in secondary schools: the Smokerface Randomized Trial: design and baseline characteristics. BMJ Open. 2016 Nov 7;6(11):e014288. doi: 10.1136/bmjopen-2016-014288. PMID 27821601
- See also: Description of the app we use. — http://www.jmir.org/2015/7/e186/